CLINICAL TRIAL: NCT04217226
Title: Evaluation of Perfusion Index-derived Parameters as Predictors of Hypotension After Induction of General Anaesthesia: a Prospective Cohort Study.
Brief Title: Perfusion Index-derived Parameters as Predictors Post-induction Hypotension.
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Bassant M. Abdelhamid, associate professor, Cairo University
Other Study IDs: MD-245-2019
Record Dates: First submitted 2020-01-02; First posted 2020-01-03 (Actual); Last update posted 2020-07-30 (Actual); Status verified 2020-07

CONDITIONS: Hypotension; General Anesthesia Induced Hypotension
MeSH Terms: conditions — Hypotension

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- study group: adult patients (18-59 years), ASA I-II-III, scheduled for elective surgeries under general anaesthesia.
  Interventions: Device: Perfusion index derived parameters

INTERVENTIONS:
Device: Perfusion index derived parameters — The PVI and PI will be recorded in the supine position by an anaesthesiologist who was not involved in the further intraoperative monitoring of the patient using Masimo SET ("MightySat 9900, Masimo Corporation, Irvine, CA, USA). This device allows bluetooth radio for transfer of parameter data to a smart device. The device will be applied on the index finger of the dominant hand of each patient. It will be applied on the hand that neither contains the venous line nor the blood pressure cuff. Three measurements of PVI and PI on one minute interval will be recorded. We will use the average of these readings.
  Dicpleth is defined as the ratio of the height of the dicrotic notch to the height of the systolic peak, measured at end-expiratory time.

SUMMARY:
The perfusion index (PI) is a numerical value for the ratio between pulsatile and non-pulsatile blood flow measured by a special pulse oximeter. PI represents the baseline sympathetic tone which is assumed one of the factors contributing for hypotension. Patients with low PI were reported by Mahendale and Rajasekhar to show greater hypotension after induction of anesthesia. This was explained by the high sympathetic tone in these patients which is suddenly masked by propofol administration leading to profound hypotension.

This study aims to evaluate the ability of preoperative plethysmographic variability index, perfusion index and the Dicrotic Plethysmography to predict post-induction hypotension.

DETAILED DESCRIPTION:
The perfusion index (PI) is a numerical value for the ratio between pulsatile and non-pulsatile blood flow measured by a special pulse oximeter. PI represents the baseline sympathetic tone which is assumed one of the factors contributing for hypotension. Patients with low PI were reported by Mahendale and Rajasekhar to show greater hypotension after induction of anesthesia. This was explained by the high sympathetic tone in these patients which is suddenly masked by propofol administration leading to profound hypotension. Moreover, The PI has been described as a reliable tool for vascular tone assessment and monitoring.

Dicrotic Plethysmography (Dicpleth): is easily derived from the photoplethysmographic signal. It represents the relative height of the dicrotic wave compared with the maximum peak of the waveform, has been described as the amount of reflected wave, dependent on the vascular tone. M.Coutrot et al quantified Dicpleth variations to detect arterial hypotension and mentioned that Dicpleth and PI are both related to vascular tone and are easily derived from the photoplethysmographic signal. Moreover, Chowienczyk PJ et. al. demonstrated that the reduction in Dicpleth is related to the reduction of vascular tone caused by vasodilator drugs, such as salbutamol or glyceryl trinitrate

ELIGIBILITY:
Inclusion Criteria:

* • Adult patients (18-59 years)

  * ASA I-II
  * Patients scheduled for elective surgeries under general anaesthesia

Exclusion Criteria:

* • Operations which will last for less than 15 minutes.

  * Patients with cardiac morbidities (impaired contractility with ejection fraction < 40% and tight valvular lesions, unstable angina).
  * Patients with heart block and arrhythmia (atrial fibrillation and frequent ventricular or supraventricular premature beat).
  * Patient with decompansted respiratory disease (poor functional capacity, generalized wheezes, peripheral O2 saturation < 90% on room air).
  * Patients with peripheral vascular disease or long standing DM affecting PVI readings.
  * Pregnancy.

Ages: 18 Years to 59 Years | Sex: All
Age Groups: Adult
Study Population: Participants will be adult patients (above 18 years), ASA I-II-III, scheduled for elective surgeries under general anaesthesia.
Sampling Method: Probability Sample
Enrollment: 93 (Actual)
Dates: Start 2020-01-20 (Actual); Primary Completion 2020-06-05 (Actual); Study Completion 2020-07-28 (Actual)

PRIMARY OUTCOMES:
The area under receiver operating characteristic (AUROC) curve for perfusion index to predict hypotension after induction of anesthesia | 10 minutes
  PI will be recorded in the supine position by an anaesthesiologist who was not involved in the further intraoperative monitoring of the patient using Masimo SET

SECONDARY OUTCOMES:
Mean arterial blood pressure | 15 minutes
  Mean arterial blood pressure will be measures in supine position in one of the upper limbs in the operating room measured at 1-minute intervals starting from preoperative baseline readings till skin incision.
Plethysmographic variability index | 10 minutes
  The area under receiver operating characteristic (AUROC) curve for Plethysmographic variability index to predict hypotension after induction of anesthesia.
Dicrotic Plethysmography | 10 minutes
  calculated as a ratio between height of the dicrotic notch to amplitude of the pulsatile component of the digital photoplethysmographic signal. The value will be obtained by averaging the values of three consecutive complexes, at end-expiratory time.
  The area under receiver operating characteristic (AUROC) curve for Dicrotic Plethysmography to predict hypotension after induction of anesthesia.
Incidence of post-induction hypotension | 15 minutes after induction of anesthesia
  defined as mean arterial pressure < 75% of the baseline reading during the period from induction of anesthesia until skin incision.
Heart rate | 5 minutes
  preoperative baseline readings
systolic arterial blood pressure | 5 minutes
  preoperative baseline readings
diastolic arterial blood pressure | 5 minutes
  preoperative baseline readings

CONTACTS AND LOCATIONS:
Overall Officials: Bassant abdelhamid, M.D., Principal Investigator — Cairo University
Locations (1):
- Anesthesia Department, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Tsuchiya M, Yamada T, Asada A. Pleth variability index predicts hypotension during anesthesia induction. Acta Anaesthesiol Scand. 2010 May;54(5):596-602. doi: 10.1111/j.1399-6576.2010.02225.x. Epub 2010 Mar 10. PMID 20236098
- [Background] Mehandale SG, Rajasekhar P. Perfusion index as a predictor of hypotension following propofol induction - A prospective observational study. Indian J Anaesth. 2017 Dec;61(12):990-995. doi: 10.4103/ija.IJA_352_17. PMID 29307905
- [Derived] Abdelhamid B, Yassin A, Ahmed A, Amin S, Abougabal A. Perfusion index-derived parameters as predictors of hypotension after induction of general anaesthesia: a prospective cohort study. Anaesthesiol Intensive Ther. 2022;54(1):34-41. doi: 10.5114/ait.2022.113956. PMID 35359139